CLINICAL TRIAL: NCT01712724
Title: Effects of Combined Resistance and Aerobic Training vs Aerobic Training on Cognition and Mobility Following Stroke
Acronym: TRI-RAvA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Ontario Stroke Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OSN1207-000144; OSN1207-000144 (Other Grant/Funding Number: OSN1207-000144)
Record Dates: First submitted 2012-10-20; First posted 2012-10-23 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Cerebrovascular Accident
Keywords: exercise therapy; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Training (Active Comparator): Walking, elliptical, stationary recumbent or upright cycling will be the modes of AT prescribed depending on individual ability and access to equipment when away from the Centre. Treadmill or overground walking will be considered for those who can sustain high enough speeds and durations to achieve aerobic benefit. Cycle ergometer exercise (upright or recumbent) will be prescribed to patients in addition to walking when stroke-related deficits preclude a sufficient walking speed. The AT group will complete AT 5 d∙wk-1.
  Interventions: Other: combined resistance and aerobic training
- Combined Resistance and Aerobic Training (Experimental): The AT+RT group will complete AT 3 d∙wk-1 + RT 2 d∙wk-1.The RT exercises will be task specific, incorporating muscle actions that are performed during daily activities. Resistance will be provided by hand-held dumbbells, exercise bands (wrist/ankle attachments), or patients' body weight. A weight load equivalent to 50-60% of 1 repetition maximum will be prescribed on the non-affected limb. On the hemiparetic limb ≥50% of 1 repetition maximum and/or a resistance rated as 13-14 on the Rating of Perceived Exertion scale on the last repetition of the set will be prescribed
  Interventions: Other: combined resistance and aerobic training

INTERVENTIONS:
Other: combined resistance and aerobic training — For the group randomized to AT+RT, Patients will gradually be progressed from 1-2 sets and then from 10-15 repetitions and then increase resistance by 1.6-5 kg or increase the exercise band level and then reduced repetitions to 10 and repeated this process.

SUMMARY:
Both aerobic training (AT) and resistance/strength training (RT) have the potential to improve recovery after stroke. Research conducted in chronic disease and healthy populations suggest that AT and RT "combination therapy" may produce synergistic and superior effects along cognition and mobility domains, when compared to AT alone. However, the effects of a combined training approach (AT+RT) compared to AT alone has not been investigated in people post-stroke.

DETAILED DESCRIPTION:
Patients referred to Toronto Rehabilitation Institute's Risk Factor Modification and Exercise Program following Stroke (TRI-REPS) will be randomized to either AT+RT or AT alone. Mobility (6 minute walk test), and cognition (Vascular Cognitive Impairment Harmonization Standards) will be measured pre- post 6 months of exercise. Secondary measures will include body composition, and biochemical changes. This project will help to determine an exercise treatment strategy that will guide best practice guidelines aimed at promoting mobility and brain health in people post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke (ischemic or hemorrhagic)
* Ability to walk at least 100 m independently with or without an assistive
* device with no severe limitations due to pain
* Living in the community at least 3 months post stroke (no upper limit)
* Stroke-related motor impairment score of 3-6 on the Chedoke-McMaster Stroke
* Assessment scale of the leg and/or foot
* Ability to provide informed consent

Exclusion Criteria:

* Unstable angina or orthostatic blood pressure decrease of > 20 mmHg
* Resting hypertension (SBP > 160 mm Hg or DBP > 100 mm Hg)
* Diabetes related or other eye/vision complications (severe proliferative retinopathy)
* Cardiovascular morbidities which would limit exercise tolerance (e.g. heart failure, hypertrophic cardiomyopathy, horizontal or downsloping ST-segment depression > 2 mm, symptomatic aortic stenosis, complex arrhythmias)
* Musculoskeletal impairments which would preclude safe participation in exercise
* Cognitive and/or behavioral issues that would significantly limit participation in exercise testing and training, prior unrelated neurological disorders or psychiatric illness
* Severe communicative aphasia or comprehensive aphasia (as noted in clinical reports)
* Patients with anxiety disorder, claustrophobia, or pacemaker implantation will be excluded from brain imaging and perfusion measures
* Exposure to a similar or identical neuropsychological battery within <6 months
* Currently smoking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 1 year
  Vascular Cognitive Impairment Harmonization Standards

SECONDARY OUTCOMES:
Body Composition | 1 year
  Fat free mass will be measured by dual energy x-ray absorptiometry
Biochemical Changes (blood samples) | 1 year
  brain-derived neurotrophic factor, insulin-like growth factor I, homocysteine, and C-reactive protein
Functional Mobility | 1 year
  Six minute walk distance

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Vanzella LM, Lawand R, Shuaib M, Oh P, Corbett D, Marzolini S. Validity of Bioelectric Impedance in Relation to Dual-Energy X-Ray Absorptiometry for Measuring Baseline and Change in Body Composition After an Exercise Program in Stroke. J Strength Cond Res. 2022 Dec 1;36(12):3273-3279. doi: 10.1519/JSC.0000000000004287. Epub 2022 Jun 1. PMID 36417356